CLINICAL TRIAL: NCT03435744
Title: A Multicentre 12-week Randomised, Double Blind, Placebo Controlled Trial of Simvastatin as Augmentation Treatment for Treatment-resistant Depression
Brief Title: Simvastatin as an Augmentation Treatment for Treatment Resistant Depression: Randomized Controlled Trial.
Acronym: DepSTAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PILL-DepSTAT-001
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: 1-Simvastatin plus TAU, 2- Placebo plus TAU
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind plcaebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin with TAU (Experimental): Participants will receive Simvastatin 20 mg added to TAU for 3 months
  Interventions: Drug: Simvastatin 20 mg
- Placebo Oral Tablet with TAU (Placebo Comparator): Participants will receive placebo added to TAU for 3 months
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Drug: Simvastatin 20 mg — Simvastatin 20 mg added to TAU for 3 months.
  Other Names: Statins
  Arms: Simvastatin with TAU
Other: Placebo Oral Tablet — Matched placebo added to TAU for 3 months
  Arms: Placebo Oral Tablet with TAU

SUMMARY:
In this double blind, randomized placebo controlled trial we aim to determine the efficacy of simvastatin as an add-on treatment for treatment resistant depression. We will recruit 150 people with treatment-resistant depression with the aim of determining whether the addition of simvastatin (20mg daily) to treatment as usual (TAU) for 12 weeks leads to an improvement in depressive symptom compared with placebo added to TAU.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 current major depressive episode
* Must currently be on an antidepressant and must have had a non-response to >2 oral antidepressant treatments in the current episode (including the one they are currently taking).
* Capacity to give informed consent
* Willing to use adequate contraception
* Give written informed consent

Exclusion Criteria:

* Primary psychotic or bipolar disorder
* History of intolerance to statins or presence of any contraindication to statins
* Presence of any serious medical condition or neurological problem
* Presence of autoimmune or inflammatory disorder
* Alcohol or drug dependence
* Active suicidal ideation
* Pregnant or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS; Montgomery Asberg, 1979) | Week-2, Week-4, Week-8 and Week-12
  The MADRS will be used as primary outcome measure in estimating depression severity

CONTACTS AND LOCATIONS:
Locations (4):
- Pakistan (4):
  - Civil Hospital, Hyderābād
  - Civil Hospital, Karachi
  - Abbasi Shaheed Hospital, Karachi
  - Institute of Professional Psychology, Rawalpindi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Husain MI, Chaudhry IB, Khoso AB, Kiran T, Khan N, Ahmad F, Hodsoll J, Husain MO, Naqvi HA, Nizami AT, Chaudhry N, Khan HA, Minhas F, Meyer JH, Ansari MA, Mulsant BH, Husain N, Young AH. Effect of Adjunctive Simvastatin on Depressive Symptoms Among Adults With Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e230147. doi: 10.1001/jamanetworkopen.2023.0147. PMID 36808239
- [Derived] Husain MI, Chaudhry IB, Khoso AB, Husain MO, Rahman RR, Hamirani MM, Hodsoll J, Carvalho AF, Husain N, Young AH. Adjunctive simvastatin for treatment-resistant depression: study protocol of a 12-week randomised controlled trial. BJPsych Open. 2019 Jan;5(1):e13. doi: 10.1192/bjo.2018.84. PMID 30762508